CLINICAL TRIAL: NCT01620203
Title: Observational Study in Preterm Infants With and Without Intracranial Hemorrhage: Longitudinal Assessment of Cerebral Oxygenation, Perfusion and Function
Brief Title: Observational Study in Preterm Infants With Intracranial Hemorrhage
Status: Completed | Type: Observational
Sponsor: Nelson Claure (Other)
Responsible Party: Sponsor-Investigator, Nelson Claure, Research Associate Professor of Pediatrics, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 20120065
Record Dates: First submitted 2012-06-05; First posted 2012-06-15 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Intracranial Hemorrhage; Intraventricular Hemorrhage; Cerebral Hypoxia
Keywords: Premature infants; Intracranial hemorrhage; Intraventricular hemorrhage; Cerebral oxygenation; Brain function; Cerebral perfusion
MeSH Terms: conditions — Intracranial Hemorrhages; Hypoxia, Brain; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Matched group of control infants without diagnosis of intracranial hemorrhage
  Interventions: Other: No intervention/treatment is given
- Intracranial Hemorrhage: Group of preterm infant with diagnosis of intracranial hemorrhage.
  Interventions: Other: No intervention/treatment is given

INTERVENTIONS:
Other: No intervention/treatment is given

SUMMARY:
Intracranial Hemorrhage (ICH) is an important morbidity affecting premature infants and can have considerable effects on neurodevelopmental outcome.

The investigators showed that preterm infants with severe ICH have decreased cerebral oxygenation several weeks after the hemorrhage. The mechanisms involved in this state of decreased cerebral oxygenation in preterm infants and the effects on cerebral function are unknown.

This longitudinal observation study will evaluate physiologic parameters to determine trends in cerebral oxygenation and function in preterm infants with ICH in comparison to infants without ICH.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 23 and 28 weeks of gestation
* Diagnosed with ICH grades II or higher during the first week after birth
* Matched control infants without ICH.

Exclusion Criteria:

* Major congenital malformations
* Birth asphyxia
* Not expected to survive

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants admitted to the newborn intensive care unit at Holtz Children's Hospital of the Jackson Memorial Hospital/University of Miami Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change in cerebral oxygenation | postnatal weeks 4 and 8
  Comparison of the progression of cerebral oxygenation measured non-invasively by near infrared spectroscopy over time in infants with ICH and non-ICH infants.

SECONDARY OUTCOMES:
Change in cerebral perfusion and function | post natal weeks 4 and 8
  Comparisons of ultrasound measurements of superior vena cava flow and brain electrical activity by electroencephalography over time in infants with ICH and non-ICH infants.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Claure, M.Sc.,Ph.D., Principal Investigator — University of Miami; Eduardo Bancalari, M.D., Principal Investigator — University of Miami; Deepak Jain, M.D., Principal Investigator — University of Miami; Sethuraman Swaminathan, M.D., Principal Investigator — University of Miami
Locations (1):
- Holtz Children's Hospital, Jackson Memorial Hospital/University of Miami Medical Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No